CLINICAL TRIAL: NCT04221750
Title: Lifestyle Intervention Plus Metformin to Treat Frailty in Older Veterans With Obesity
Brief Title: Diet and Exercise Plus Metformin to Treat Frailty in Obese Seniors
Acronym: DEMFOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Michael E. DeBakey VA Medical Center (U.S. Federal Agency); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENDA-007-19F; H-46970 (Other Grant/Funding Number: VA Office of Research and Development)
Record Dates: First submitted 2020-01-02; First posted 2020-01-09 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Frailty; Sarcopenic Obesity; Aging
MeSH Terms: conditions — Frailty | interventions — Exercise; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lifestyle Therapy plus Metformin (Experimental): Diet-induced weight loss and Exercise Training plus Metformin 1500 mg daily
  Interventions: Behavioral: Lifestyle therapy; Drug: Metformin Hydrochloride
- Lifestyle Therapy plus Placebo (Placebo Comparator): Diet-induced weight loss and Exercise Training plus Placebo
  Interventions: Behavioral: Lifestyle therapy; Drug: Placebo
- Healthy lifestyle plus Metformin (Active Comparator): Healthy lifestyle and Metformin 1500 mg daily
  Interventions: Drug: Metformin Hydrochloride; Behavioral: Healthy Lifestyle

INTERVENTIONS:
Behavioral: Lifestyle therapy — Weight management program, in which participants are prescribed a balanced diet that provides and energy deficit of 500 to 750 kcal per day to induced ~10% weight loss plus Supervised combined aerobic and resistance exercise training three times weekly
  Other Names: Diet-induced weight loss and exercise training
  Arms: Lifestyle Therapy plus Metformin; Lifestyle Therapy plus Placebo
Drug: Metformin Hydrochloride — Given orally starting at 500 mg (one tablet) taken orally once a day with meals. After a week, the dose of metformin will be increased to 1000 mg (two tablets) daily. After another week, the dose of metformin will be increased to 1500 mg (three tablets) daily.
  Arms: Healthy lifestyle plus Metformin; Lifestyle Therapy plus Metformin
Drug: Placebo — Given orally starting at 500 mg (one tablet) taken orally once a day with meals. After a week, the dose of placebo will be increased to 1000 mg (two tablets) daily. After another week, the dose of placebo will be increased to 1500 mg (three tablets) daily.
  Arms: Lifestyle Therapy plus Placebo
Behavioral: Healthy Lifestyle — Group educational sessions that focus on healthy diet, exercise, and social support once a month
  Arms: Healthy lifestyle plus Metformin

SUMMARY:
The continuing increase in prevalence of obesity in older adults including many older Veterans has become a major health concern. The clinical trial will test the central hypothesis that a multicomponent intervention consisting of lifestyle therapy (diet-induced weight loss and exercise training) plus metformin will be the most effective strategy for reversing sarcopenic obesity and frailty in older Veterans with obesity.

DETAILED DESCRIPTION:
The growing prevalence of obesity in older adults including many older Veterans, has become a major concern in the US already strained health care system in general and in the VA in particular. In older adults, obesity exacerbates the age-related decline in physical function resulting in frailty, decrease in quality of life, loss of independence, and increase in nursing home admissions. The investigators' group demonstrated that weight loss from lifestyle therapy improves physical function and ameliorates frailty but the improvement was modest at best and most obese older adults remained frail. More importantly, there are concerns that the weight-loss induced loss of muscle and bone mass could worsen underlying age-related sarcopenia and osteopenia in the subset of frail obese elderly. Metformin, a biguanide, is a widely available drug used as first line treatment of type 2 diabetes. Animal studies suggest that metformin improves health span and increases lifespan, hence may represent a novel intervention for frailty. Because metformin reduces cellular senescence and senescence-associated phenotype (SASP), it is believed to retard accelerated aging most especially in older adults with obesity. The objective is to conduct a head-head comparative efficacy, placebo controlled, randomized controlled trial to test the hypothesis that lifestyle therapy + metformin for six months will be more effective than lifestyle therapy alone or metformin alone in improving physical function and preventing the weight loss-induced reduction in muscle and bone mass in obese (BMI > 30 kg/m2) older (age 65 - 85 years) Veterans with physical frailty.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 - 85 years
* BMI = or > 30 kg/m2
* Mild to moderate frailty (score of 18 to 31 in the modified Physical Performance Test)
* Stable body weight (plus/minus 2 kg) during the past 6 months
* Sedentary (regular exercise <1 h/wk or <2 x/wk for the last 6 months)
* Willing to provide informed consent

Exclusion Criteria:

* Any major chronic diseases, or any condition that would interfere with exercise or dietary restriction, or use of metformin, in which exercise, dietary restrictions, or metformin are contraindicated, or that would interfere with interpretation of results
* Cardiopulmonary disease (e.g. recent MI, unstable angina, stroke) or unstable disease (e.g., NYHA Class III or IV congestive heart failure, severe pulmonary disease requiring steroid pills or the use of supplemental oxygen) that would contraindicate exercise or dietary restriction
* Severe orthopedic (e.g. awaiting joint replacement) and/or neuromuscular (e.g. multiple sclerosis, active rheumatoid arthritis) disease or impairments that would contraindicate participation in exercise
* Renal impairment as defined by an estimated glomerular filtration rate (eGFR of less than 30 mL/min/1.73 m2) in which metformin is contraindicated
* Other significant co-morbid disease that would impair ability to participate in the exercise intervention (e.g. severe psychiatric disorder [e.g. bipolar, schizophrenia], excess alcohol use [>14 drinks per week])
* Severe visual or hearing impairments that would interfere with following directions
* Significant cognitive impairment, defined as a known diagnosis of dementia or positive screening test for dementia using the Mini-Mental State Exam (i.e. MMSE score <24)69
* Uncontrolled hypertension (BP>160/90 mm Hg)
* History of malignancy during the past 5 years (except non-melanoma skin cancers)
* Current use of bone acting drugs (e.g. use of estrogen, or androgen containing compound,raloxifene, calcitonin, parathyroid hormone during the past year or bisphosphonates during the last two years)
* Osteoporosis (T-score -2.5 and below on hip or spine scan) or history of fragility fractures
* Known history of diabetes mellitus or any of the following:
* Fasting blood glucose of 126 mg/dl, or HbA1c of 6.5% or >
* Terminal illness with life expectancy less than 12 months, as determined by a physician
* Use of any drugs or natural products designed to induce weight loss within past three months
* History of excessive alcohol consumption (e.g. 8 or more drinks a week for women and 15 or more drinks a week for men)
* Positive exercise stress test for ischemia or any indication for early termination of exercise stress testing
* Taking metformin or any other glucose lowering drug
* Lives outside of the study site or is planning to move out of the area in the next 2 years

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 114 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Change in the modified Physical Performance Test (PPT) | 6 months
  The Physical Performance Test includes seven standardized tasks (walking 15.2 m [50 ft], putting on and removing a coat, picking up a penny, standing up from a chair, lifting a book, climbing one flight of stairs, and performing a progressive Romberg test) plus two additional tasks (going up and down four flights of stairs and making a 360-degree turn). The score for each task ranges from 0 to 4, with higher scores indicating better physical performance; a perfect score would be 36.

SECONDARY OUTCOMES:
Change in muscle strength | 6 months
  Assessed by biodex dynamometer and1-repetition maximum
Change in gait speed | 6 months
  Assessed by time need to walk a certain distance
Change in peak aerobic power | 6 months
  Assessed by indirect calorimetry during a graded exercise test
Change in lean body mass | 6 months
  Assessed by dual-energy x-ray absorptiometry (DXA)
Chang in body fat | 6 months
  Assessed by DXA
Change in thigh muscle | 6 months
  Assessed by magnetic resonance imaging (MRI)
Change in bone microarchitecture | 6 months
  Assessed by high-resolution peripheral quantitative computed tomograph (HR-pQCT)
Change in bone strength | 6 months
  Assessed by finite-element analyses
Change in hip, lumbar spine, and wrist bone mineral density (BMD) | 6 months
  Assessed by DXA
Change in serum C-telopeptide | 6 months
  Assessed by immunoassay
Change in telomere length | 6 months
  Assessed by Q-PCR
Change in mood | 6 months
  Assessed by geriatric depression scale (score range: 0 to 30, where lower scores indicating better mood)
Change in serum procollagen type 1 N propeptide | 6 months
  Assessed by radioimmunoassay
Change in serum 25-OH vitamin D | 6 months
  Assessed by immunoassay
Change in serum parathyroid hormone | 6 months
  Assessed by immunoassay
Change in high-sensitivity c-reactive protein | 6 months
  Assessed by immunoassay
Change in p16 and other markers of cell arrest | 6 months
  Assessed by immunohistochemistry
Change in protein expression of senescence associated secretory phenotype | 6 months
  Assessed by elisa or western blotting
Change in Medical Outcomes 36-Item short form Health survey (SF-36) | 6 months
  Assessed by Physical component summary and mental component summary score (score range 0 to 100, with higher scores indicating better health status)
Change in Impact of Weight on Quality of Life_Lite (IWQOL-lite) score | 6 months
  Assessed by IWQO-liteL questionnaire
Change in serum adiponectin | 6 months
  Assessed by ELISA
Change in serum leptin | 6 months
  Assessed by ELISA
Change in fasting serum insulin | 6 months
  Assessed by immunoassay
Change in fasting serum glucose | 6 months
  Assessed by glucose oxidase method
Change in blood pressure | 6 months
  Assessed by sphygmomanometry
Change in serum lipids | 6 months
  Assessed by automated enzymatic/colorimetric assays
Change in insulin growth factor 1 | 6 months
  Assessed by immunoassay
Change in Cognitive composite scores | 6 months
  Using cognitive toolbox which yields the following summary scores: Cognitive Function
  Composite Score, Fluid Cognition Composite Score, and Crystallized Cognition Composite Score (score range: -3 to +3 for each with higher scores indicating better cognitive status

CONTACTS AND LOCATIONS:
Overall Officials: Dennis T Villareal, MD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Publications from this research will be made available to the public through the National Library of Medicine PubMed Central website within one year after the date of publication (guidance is provided on the ORD website).
  MEDVAMC will not provide unrestricted, open public access to large scale health related datasets because of re-identification concerns and the obligation to protect Veterans' private information. However, controlled public access will be provided to the greatest extent possible under specific DUAs or other written agreements, and open access will be provided to the final datasets underlying peer-reviewed publications (aggregated data that can be released with privacy and confidentiality risks).

DOCUMENTS (1):
  • Informed Consent Form (2024-09-13): https://cdn.clinicaltrials.gov/large-docs/50/NCT04221750/ICF_000.pdf